CLINICAL TRIAL: NCT00681603
Title: The Application of Subconjunctival Injection of Bevacizumab (Avastin) in the Treatment of Corneal Neovasculization
Brief Title: Safety and Effectiveness of Subconjunctival Injection of Bevacizumab in the Treatment of Corneal Neovasculization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wei-Li Chen/Assistant Professor, National Taiwan University, Department of Ophthalmology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200708015M
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2007-08

CONDITIONS: Lipid Keratopathy; Penetrating Keratoplasty; Herpetic Keratopathy; Rosacea
Keywords: corneal neovascularization; lipid keratopathy; penetrating keratopathy; bevacizumab; Avastin; subconjunctival injection
MeSH Terms: conditions — Rosacea; Corneal Neovascularization | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): 13 cases that accepted subconjunctival injection of bevacizumab
  Interventions: Drug: subconjunctival injection of bevacizumab ( 1.25 to 2.50 mg)

INTERVENTIONS:
Drug: subconjunctival injection of bevacizumab ( 1.25 to 2.50 mg) — subconjunctival injection of bevacizumab ( 1.25 to 2.50mg) according to the clinical judgment. Once per months for three times then reevaluate the drug effect, if the response was adequate, stop the trial; if no improvement, another three month intervention would be performed.
  Other Names: bevacizumab ( Avastin )

SUMMARY:
1. Purpose:Our animal study demonstrated the effectiveness of subconjunctival injection of bevacizumab in the inhibition of corneal neovasculization formation. The purpose of this human interventional study is to report the treatment outcome of subconjunctival injection of bevacizumab in patients with corneal neovascularization.
2. Material and methods: We enrolled 13 patients with unilateral or bilateral clinically significant corneal neovascularization during Aug. 2007 to Jan. 2008. Subconjunctival injection of bevacizumab once per month for at most 7 times was performed according to clinical response.
3. Main outcome measurements: resolution of corneal neovascularization, reduction of lipid infiltrate, improved visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Significant unilateral or bilateral corneal neovascularization that extending over the limbus at least 2mm
* The underlying etiologies that caused corneal neovascularization included post penetrating keratoplasty (PKP), trauma, infectious or non-infectious corneal ulcer, post-keratoplasty, etc.
* Corneal neovascularization induced lipid keratopathy, corneal edema, or irregular corneal surface. The best-corrected visual acuity was less than 20/25
* Post-PKP corneal neovascularization that had no associated lipid keratopathy, no corneal edema, or corneal irregularity. But the neovascularization was highly possible to cause graft rejection.
* The corneal neovascularization was refractory to other medical treatment
* The patient had received PKP or other corneal surgeries more than half a year ago and was not in the acute post-operation phase
* The patient had no active endopthalmitis, glaucoma with uncontrolled intraocular pressure, or vitreoretinal diseases
* The patient signed inform consent to have regular follow up and treatment

Exclusion Criteria:

* The neovascularization had clinical improvement three months before the first injection
* The lipid keratopathy had clinical improvement three months before the first injection
* The patient that suspected to have poor visual outcome or had already been light sense negative
* Glaucoma patient that had uncontrolled intraocular pressure
* Poor corneal epithelialization
* Post-PKP patient that had graft failure or rejection
* Patient that had systemic disease which was not suitable for bevacizumab use
* Pregnant patient

Ages: 10 Years to 70 Years | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Resolution of corneal neovascularization, reduction of lipid infiltrate, improved visual acuity | prospective

SECONDARY OUTCOMES:
major side effects | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Ophthalmology, National Taiwan University Hospital,, Taipei, Taipei, Taiwan